CLINICAL TRIAL: NCT03463876
Title: A Phase II, Single-arm, Open-labeled Trial of SHR-1210 (an Anti-PD-1 Inhibitor) in Combination With Apatinib in Patients With Advanced HCC
Brief Title: A Trial of SHR-1210 (an Anti-PD-1 Inhibitor) in Combination With Apatinib in Patients With Advanced HCC(RESCUE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-APTN-Ⅱ-208-HCC
Record Dates: First submitted 2018-03-07; First posted 2018-03-13 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2022-06

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1210+Apatinib (Experimental): Patients will received apatinib orally every day and SHR-1210 200mg (3mg/kg for underweight patients) iv every 2 weeks.
  Interventions: Drug: SHR 1210+apatinib

INTERVENTIONS:
Drug: SHR 1210+apatinib — SHR-1210 200mg (3mg/kg for underweight patients) iv every 2 weeks;Apatinib,250 mg/day.

SUMMARY:
The purpose of this study is to observe and preliminary explore the efficacy and safety of combination of Apatinib and SHR-1210 regimen in treating advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
SHR-1210 is a humanized monoclonal antibody against Programmed death 1(PD-1). Apatinib is a new kind of selective Vascular Endothelial Growth Factor Receptor 2(VEGFR-2) tyrosine kinase inhibitor (TKI).

Patients with advanced HCC who failed or intolerable to sorafenib will received apatinib 250mg orally every day and SHR-1210 200mg (3mg/kg for underweight patients) iv every 2 weeks. The efficacy and safety will be observed.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years old, both genders.
2. Conform to the clinical diagnosis standard strictly or histological or cytological confirmation of HCC(hepatocellular carcinoma) and with at least one measurable lesion by computed tomography (CT) scan or magnetic resonance imaging (MRI) according to RECIST 1.1.
3. Liver function status Child-Pugh Class A.
4. Barcelona Clinic Liver Cancer stage Category B or C.
5. Failure or intolerance to prior treatment with targeted therapy.
6. Eastern Cooperative Oncology Group Performance Status of 0 or 1.
7. Life expectancy of at least 12 weeks.
8. Adequate bone marrow, liver and renal function (without blood transfusion, without growth factor or blood components support within 14 days before enrollment).

Exclusion Criteria:

1. Patients with any active autoimmune disease or history of autoimmune disease, including but not limited to the following: hepatitis, pneumonitis, uveitis, colitis (inflammatory bowel disease), hypophysitis, vasculitis, nephritis, hyperthyroidism, and hypothyroidism, except for subjects with vitiligo or resolved childhood asthma/atopy. Asthma that requires intermittent use of bronchodilators or other medical intervention should also be excluded.
2. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids. Doses > 10 mg/day prednisone or equivalent are prohibited within 2 weeks before study drug administration.
3. More than one regimen.
4. Known history of hypersensitivity to any components of the SHR-1210 formulation, or other antibody formulation.
5. Known or occurrence of central nervous system (CNS) metastases or hepatic encephalopathy.
6. Patients with tumor burden ≥50% of the liver volume or received liver transplantation.
7. Patients with clinical symptoms of ascites.
8. Hypertension and unable to be controlled within normal level following treatment of anti-hypertension agents(within 3 months): systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg.
9. Clinically significant cardiovascular and cerebrovascular diseases, including but not limited to severe acute myocardial infarction within 6 months before enrollment, unstable or severe angina, or coronary artery bypass surgery, Congestive heart failure (New York heart association (NYHA) class > 2), ventricular arrhythmia which need medical intervention.
10. Coagulation abnormalities (INR>2.0、PT>16s), with bleeding tendency or are receiving thrombolytic or anticoagulant therapy.
11. Previous digestive tract bleeding history within 3 months or evident gastrointestinal bleeding tendency, such as: esophageal varices, local active ulcerative lesions, gastric ulcer and duodenal ulcer, the ulcerous colitis, gastrointestinal diseases such as portal hypertension or resection of tumor with bleeding risk, etc.
12. Previous Arterial/venous thrombosis events within 3 months.
13. Proteinuria ≥ (++) and 24 hours total urine protein > 1.0 g.
14. Prior systemic chemotherapy, radiotherapy, immunotherapy, hormone therapy, surgery or target therapy within 4 weeks (Or 5 half-life of the drug, calculate the longer ) before the study drug administration, or any unresolved AEs > Common Terminology Criteria for Adverse Events (CTCAE) Grade 1.
15. Active infection or an unexplained fever > 38.5°C during screening visits or on the first scheduled day of dosing.
16. History of immunodeficiency or human immunodeficiency virus (HIV) infection.
17. HBV DNA>2000 IU/ml（or 104copies/ml），HCV RNA>103copies/ml，HBsAg+ and anti-HCV+；
18. Patients with other malignant tumor (except cured skin basal cell carcinoma and cervical carcinoma).
19. Patients who has bone metastasis, has received Palliative radiotherapy (radiotherapy area > 5% marrow area).
20. Patients must not have had prior treatment with SHR-1210 or any other PD-L1 or PD-1 antagonists or apatinib.
21. Patients who may receive live vaccine during the study, or previous had vaccination within 4 weeks.
22. Any other medical, psychiatric, or social condition deemed by the investigator to be likely to interfere with a subject's rights, safety, welfare, or ability to sign informed consent, cooperate, and participate in the study or would interfere with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 12 months
  Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).

SECONDARY OUTCOMES:
Duration of Response (DoR) | Up to approximately 12 months
  Duration of Response (DoR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
Disease Control Rate (DCR) | Up to approximately 12 months
  Disease Control Rate (DCR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
Time to objective response(TTR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1). | Up to approximately 12 months
  Time to objective response，TTR
9-month survival rate | Up to approximately 12 months
  9-month survival rate
12-month survival rate | Up to approximately 12 months
  12-month survival rate
Overall survival(OS) | Up to approximately 18 months
  Overall survival(OS)
Progression-free survival(PFS) | Up to approximately 12 months
  Progression-free survival(PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of the Chinese Academy of Military Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhou X, Cao J, Topatana W, Xie T, Chen T, Hu J, Li S, Juengpanic S, Lu Z, Zhang B, Wang K, Feng X, Shen J, Chen M. Evaluation of PD-L1 as a biomarker for immunotherapy for hepatocellular carcinoma: systematic review and meta-analysis. Immunotherapy. 2023 Apr;15(5):353-365. doi: 10.2217/imt-2022-0168. Epub 2023 Feb 27. PMID 36852452
- [Derived] Xu J, Shen J, Gu S, Zhang Y, Wu L, Wu J, Shao G, Zhang Y, Xu L, Yin T, Liu J, Ren Z, Xiong J, Mao X, Zhang L, Yang J, Li L, Chen X, Wang Z, Gu K, Chen X, Pan Z, Ma K, Zhou X, Yu Z, Li E, Yin G, Zhang X, Wang S, Wang Q. Camrelizumab in Combination with Apatinib in Patients with Advanced Hepatocellular Carcinoma (RESCUE): A Nonrandomized, Open-label, Phase II Trial. Clin Cancer Res. 2021 Feb 15;27(4):1003-1011. doi: 10.1158/1078-0432.CCR-20-2571. Epub 2020 Oct 21. PMID 33087333